CLINICAL TRIAL: NCT05960786
Title: Treating the Symptoms of Vertigo in a Real-world Setting Using the OtoBand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otolith Labs (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLith10702
Record Dates: First submitted 2023-05-18; First posted 2023-07-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Vertigo; BPPV; Meniere Disease; Labrynthitis; Vestibular Disorder; Vestibular Migraine; Benign Paroxysmal Positional Vertigo; Ménière's Vertigo; Migraine Associated Vertigo; Uncompensated Unilateral Vestibulopathy
MeSH Terms: conditions — Vertigo; Meniere Disease; Vestibular Diseases; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- 1. Moderate or Worse (MoW) Arm (Experimental): Participants will be randomized to use the Otoband as instructed by clinical coordinator per study protocol. There are 4 power levels, these participants will receive the experimental device.
  Interventions: Device: Otoband Experimental
- 2. Moderate or Worse (MoW) Arm (Sham Comparator): Participants will be randomized to use the Otoband as instructed by clinical coordinator per study protocol. There are 4 power levels, these participants will receive the sham device.
  Interventions: Device: Otoband Sham
- 1. Quality of Life (QoL) Arm (Experimental): Participants will be randomized to use the Otoband as instructed by clinical coordinator per study protocol. There are 4 power levels, these participants will receive the experimental device.
  Interventions: Device: Otoband Experimental
- 2. Quality of Life (QoL) Arm (Sham Comparator): Participants will be randomized to use the Otoband as instructed by clinical coordinator per study protocol. There are 4 power levels, these participants will receive the sham device.
  Interventions: Device: Otoband Sham

INTERVENTIONS:
Device: Otoband Experimental — Participants will be randomly assigned to use the Otoband to determine effectiveness in providing temporary relief to symptoms of vertigo.
  Arms: 1. Moderate or Worse (MoW) Arm; 1. Quality of Life (QoL) Arm
Device: Otoband Sham — Participants will be randomly assigned to use the Otoband sham to determine effectiveness in providing temporary relief to symptoms of vertigo.
  Arms: 2. Moderate or Worse (MoW) Arm; 2. Quality of Life (QoL) Arm

SUMMARY:
The goal of this virtual clinical trial is to determine the effectiveness of two study devices in providing temporary relief to adults aged 18-70 who suffer from symptoms of chronic vestibular vertigo.

The main question[s] it aims to answer are:

* Within an episode, is there a significant difference between the randomized study devices at the individual timepoints during the vertigo episode?
* Within an episode, is there evidence of quantitative treatment at each individual timepoint during the vertigo episode?

Participants will be:

* Enrolled up to 49 days; 14 days in Baseline Phase (no device) and 21 days in Treatment Phase (study device) for Study Arm 1 or 28 days in Treatment Phase (study device) for Study Arm 2
* Randomized and stratified into groups based on diagnosis to be assigned a study device
* Asked to use the study device as instructed by the study coordinator
* Asked to download a study app to submit daily diaries regarding their symptoms and use of device, and to participate in tele-health visits with study coordinators
* Asked to provide their vertigo diagnosis from their physician
* Compensated for their participation

Researchers will compare the randomized groups to see which groups respond better to which device.

DETAILED DESCRIPTION:
This study is decentralized clinical trial. This study uses technology and and virtual meetings to communicate with study participants and collect study data. This study seeks to enroll until 36 participants in the Moderate or Worse (MoW) arm have completed the study, and until 72 participants have completed the Quality of Life (QoL) arm.

All study participants that meet all of the inclusion, none of the exclusion criteria, and sign informed consent will be enrolled in the study. Participants will complete a one day enrollment meeting and an approximately 14 day Baseline Phase.

After the Baseline Phase, participants will be placed in one of two groups Moderate or Worse (MoW) group or Quality of Life (QoL) group based on the data collected about their vertigo during the Baseline Phase.

Participants will then be randomized within their assigned group (MoW or QoL) at a 2:1 ratio to an active arm or sham arm to begin the Treatment Phase of the study. Participants will be sent a study device to use when they have a vertigo episode.

Participants that enroll in the study are expected to participate up to 49 days with virtual meetings at the approximate intervals:

MoW Group: Day 4, Day 16, Day 21, Day 24, Day 31, and Day 42 QoL Group : Day 4, Day 16, Day, 21, Day 24, Day 31, and Day 49

Participants will be required to complete the DHI (Dizziness Handicap Index), VSS (Vertigo Symptom Scale), Global Impression of Symptoms, and Global Impression of Change questionnaires.

Otolith Labs received Therapeutic Breakthrough Device designation by the FDA in May 2021.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, an individual must meet all the following criteria:

  * Diagnosed as having vestibular vertigo that is caused by one or more of:

    * Benign paroxysmal positional vertigo (BPPV)
    * Migraine associated vertigo (MAV, aka vertiginous migraines)
    * Meniere's disease (aka idiopathic endolymphatic hydrops)
    * Uncompensated unilateral vestibulopathy (such as arising from vestibular neuritis and labyrinthitis)
  * Vertigo that has been present for at least 90 days
  * Score greater than 35, and less than 91, on the Dizziness Handicap Inventory (corresponding to moderate to severe vertigo)
  * Smartphone, computer or tablet and access to internet for online enrollment, check-in and wrap-up meetings
  * Willingness to install and use the JotForm ePRO app
  * Residing in the United States
  * Willingness to be paid via Venmo or PayPal.

Exclusion Criteria:

* Surgery to the base of the skull within the last 6 months or plans for surgery to the skull during enrollment period
* Any skull or neck implants such as but not limited to a cochlear implant, vascular stents, bone conduction implant, or deep brain stimulation device
* History of vitreous detachment (aka floaters) in the last 90 days
* Superior canal dehiscence (aka third window) or otic capsule dehiscence
* Hyperacusis (aka hypersensitivity to loud sounds)
* Currently undergoing vestibular rehabilitation therapy or planning to start vestibular rehabilitation therapy during the study. (People who have completed vestibular rehabilitation therapy, but in whom vestibular vertigo persists, will be permitted to enroll)
* History of cerebrovascular disorders
* Posterior fossa tumors (brain tumors located in the caudal third of the skull)
* Vestibular schwannoma (non-cancerous tumor located on the vestibulo-cochlear nerve)
* Cerebellar degeneration (progressive worsening of neurons behind the brain stem)
* Taking benzodiazepines (e.g., clonazepam, lorazepam, diazepam) for vestibular issues.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Moderate or Worse Change in Vertigo Severity | Through 21 days of treatment phase of "moderate of worse" arm of study
  Change in participant response to "How severe is your vertigo right now?" during vertigo episodes, compared to responses in baseline phase
Quality of Life Change in Scores | Day 28 of treatment phase of "quality of life" arm of study
  Change in participant's Vertigo Symptom Scale (VSS) score, compared to baseline VSS score

SECONDARY OUTCOMES:
Device Effectiveness | 30 minutes post vertigo episode during the treatment phase
  Percent change in mean severity of vertigo episodes as reported by the participant during the Treatment phase, compared to the Baseline phase.

OTHER OUTCOMES:
Effectiveness of Rating Scales | Through 21 days of treatment phase of "moderate of worse" arm of study
  Comparison of Verbal Rating Scale vs. Numerical Rating Scale as representation of participant response to device treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Principal Investigator — Otolith Labs
Locations (1):
- Otolith Labs, Washington D.C., District of Columbia, United States